CLINICAL TRIAL: NCT06702228
Title: Precision Diagnosis and Care for Families With Pulmonary Fibrosis in Ireland [PRECISE-PF]
Brief Title: Precision Diagnosis and Care for Families With Pulmonary Fibrosis in Ireland
Acronym: PRECISE-PF
Status: Recruiting | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: patientMpower Ltd. (Industry); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: PRECISE-PF
Record Dates: First submitted 2024-06-06; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-06

CONDITIONS: Connective Tissue Diseases; Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Familial Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Pulmonary Fibrosis Interstitial
Keywords: Genetic diseases; Diagnosis, Computer-assisted; Early Diagnosis; Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias
MeSH Terms: conditions — Connective Tissue Diseases; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Genetic Diseases, Inborn; Disease; Idiopathic Interstitial Pneumonias | interventions — Walk Test; Genetic Testing; Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, plasma, serum, white blood cells, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Familial pulmonary fibrosis group: Patients meeting the study inclusion criteria with an multidisciplinary team (MDT) diagnosis of a fibrotic interstitial lung disease, reporting one or more relatives with a fibrotic form of ILD
  Interventions: Diagnostic Test: Six minute walk test (6MWT); Diagnostic Test: Computer-tomography of the thorax (CT Thorax); Other: Quality of life questionnaires.; Diagnostic Test: Genetic Testing; Diagnostic Test: Spirometry; Diagnostic Test: Serology; Other: PatientMPower Home Monitoring App
- Idiopathic pulmonary fibrosis group: Patients meeting the study inclusion criteria with an MDT diagnosis of IPF in accordance with consensus criteria, ATS, ERS, JRS, ALAT guidelines, without a family history of pulmonary fibrosis.
  Interventions: Diagnostic Test: Six minute walk test (6MWT); Diagnostic Test: Computer-tomography of the thorax (CT Thorax); Other: Quality of life questionnaires.; Diagnostic Test: Genetic Testing; Diagnostic Test: Spirometry; Diagnostic Test: Serology; Other: PatientMPower Home Monitoring App
- Connective tissue disease related interstitial lung disease group: Patients meeting the study inclusion criteria who meet the American College of Rheumatology/European League Against Rheumatism criteria for rheumatoid arthritis, scleroderma, Sjogren's syndrome, idiopathic inflammatory myopathy and systemic lupus erythematosus criteria
  Interventions: Diagnostic Test: Six minute walk test (6MWT); Diagnostic Test: Computer-tomography of the thorax (CT Thorax); Other: Quality of life questionnaires.; Diagnostic Test: Genetic Testing; Diagnostic Test: Spirometry; Diagnostic Test: Serology; Other: Other Quality of Life Questionnaires; Other: PatientMPower Home Monitoring App

INTERVENTIONS:
Diagnostic Test: Six minute walk test (6MWT) — Assessment of exercise capacity by the carrying out of a 6MWT at 0, 6 and 12 months.
Diagnostic Test: Computer-tomography of the thorax (CT Thorax) — Radiological assessment via CT Thorax, preferably high-resolution CT thorax at baseline on entering the study and at one year. CT images will be collected on study end. CT images in all subjects will be evaluated by three readers blinded to any other interpretation and conforming to ATS-guidelines. Coded data from CT scans will be shared with our collaborator Professor Simon Walsh at Imperial College, London who will use computational methods to identify novel radiologic phenotypes linked to disease behaviour of our patient's fibrotic lung disease.
Other: Quality of life questionnaires. — Qality of life questionnaires including; modified Medical Research Council (mMRC) dyspnea scale, The King's Brief Interstitial Lung Disease Questionnaire (KBILD), The Leister Cough Questionnaire and the EQ-5D-3L questionnaire are measured at 0, 6 and 12 months
Diagnostic Test: Genetic Testing — 10ml of serum will be collected for DNA extraction and analysed for causative and at risk genetic mutations
Diagnostic Test: Spirometry — We will carry out spirometry at baseline, 6 and 2 months including forced vital capacity and diffusing capacity of the lungs for carbon monoxide.
Diagnostic Test: Serology — Serology which may indicate an underlying diagnosis of ILD will be carried out on study entry. This will include a full blood count, renal profile, liver profile, C-reactive protein, creatine kinase, erythrocyte sedimentation rate, antinuclear antibodies, anticyclic citrullinated peptide antibodies, rheumatoid factor, an extended myositis antibody panel, sjögren's antibodies, scleroderma antibodies and a hypersensivity pneumonitis panel if clinically indicated.
Other: Other Quality of Life Questionnaires — Patient Global Assessment and Clinician Global Assessment scores completed at 0, 6 and 12 months
  Groups: Connective tissue disease related interstitial lung disease group
Other: PatientMPower Home Monitoring App — Continuous at home monitoring of patients using home-based digital spirometry and pulse-oximetry with real-time feedback readings to patient and clinician. Smartphone app for patients, spirometer and pulse oximeter are connected to the app via Bluetooth. Patients are asked to take 2 readings per week.

SUMMARY:
This study aims to improve the understanding of how genes and the environment can influence and cause pulmonary fibrosis. By identifying the presence of genes and other factors that can put people at risk of developing pulmonary fibrosis, the influence these factors have on the progression of the disease can be studied.

Interstitial lung disease (ILD) is the medical term given to a group of lung diseases affecting the same part of the lung, the interstitium, each with similar symptoms. In some of these diseases, inflammation leads to lung scarring, known as fibrosis. Idiopathic Pulmonary Fibrosis (IPF) is one of these diseases; it has a particular pattern on computed tomography (CT) scans. IPF is 'idiopathic' as it is not yet fully understood why it happens. It has a poor prognosis. The average survival time is three to five years after diagnosis. While new antifibrotic drugs offer hope of slowing disease progression, lung transplant is the only cure, and it comes with its significant risks.

Although it is not fully understood what causes IPF, it is known that genetic factors significantly increase the risk of developing the disease. Up to a quarter (25%) of people with IPF with a family history appear to have a causative genetic variant. Familial-pulmonary-fibrosis (FPF), the term for people with at least one relative with IPF, may have worse disease when compared to those without a family history. However, this needs more research. Patients with specific genes, telomere-related gene variants, appear to have a greater risk of developing blood disorders from medications given to suppress the body's immune system after a lung transplant.

Progressive pulmonary fibrosis is pulmonary fibrosis where there is irreversible worsening of the disease, worsening of lung function, respiratory symptoms and even early death. It is of growing importance regardless of the cause, whether it be idiopathic, familial or secondary to a connective tissue disease. ILD is increasingly recognised as a complication of connective tissue diseases. It is the leading cause of death in people with systemic sclerosis. The new antifibrotic drugs slow the progression of CTD-ILD. People with progressive pulmonary fibrosis who have a greater than 10% drop over one year in a measure of their lung function, called the forced vital capacity, benefit most from antifibrotic therapy. Early identification of people with progressive disease would allow the commencement of treatment quicker. At-home spirometry may be a way of identifying those who are worsening early.

This study hypothesises that by improving knowledge of factors that affect disease behaviour and progression and assessing tools for the early identification of progressive disease, such as at-home spirometry and CT scan pattern determination by deep-learning analysis, we can provide 'precision' diagnosis and treatment. It is hoped that this improved understanding will help reduce the clinical risk for people with pulmonary fibrosis and their families.

This study aims to recruit 300 patients: 100 with IPF, 100 with FPF, and 100 with CTD ILD. Each participant will be followed for one year.

This observational study aims to help answer a number of questions:

1. What genetic variants cause people to develop ILD, and which increase a person's risk of developing ILD are present in the study population?
2. How does pulmonary fibrosis behave in people who have a family history of IPF compared to those who do not and in people with CTD-ILD?
3. Are different types of pulmonary fibrosis more progressive than others i.e. Is pulmonary fibrosis in those with a family history of pulmonary fibrosis more progressive than in those who do not have a family history?
4. Is the disease in those with a genetic variant known to cause ILD worse than in those who don't have a gene?
5. Can at-home spirometry help identify people at risk of progressive disease early?
6. Can deep-learning analysis (AI) be used to find CT scan patterns to predict when pulmonary fibrosis will worsen?

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* An MDT diagnosis of fibrotic ILD which fall into one of the following three catagories;

  1. Have a multidisciplinary team (MDT) diagnosis of a fibrotic interstitial lung disease, reporting one or more relatives with a fibrotic form of ILD
  2. Have a MDT diagnosis of IPF in accordance with consensus criteria, ATS, ERS, JRS, ALAT guidelines without a family history of pulmonary fibrosis.
  3. Meet the American College of Rheumatology/European League Against Rheumatism criteria for rheumatoid arthritis, scleroderma, Sjogren's syndrome, idiopathic inflammatory myopathy and systemic lupus erythematosus.

Exclusion Criteria:

* Currently participating in an interventional clinic trial.
* Change in clinical phenotype from initial radiological diagnosis to screening.
* Acute or chronic hypersensitivity pneumonitis with consensus criteria (appropriate exposure history, radiological features ± avian and fungal precipitins).
* Asbestosis (appropriate occupational history and radiological evidence of asbestos exposure)
* Life expectancy for any disease, including ILD <12 months (investigator assessment)
* Major extrapulmonary physiological restriction (e.g. chest wall abnormality, large pleural effusion)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who meet the study criteria will be recruited from the rheumatology and respiratory clinics in Beaumont Hospital, a tertiary hospital in Dublin, Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Determine if familial-pulmonary-fibrosis is more progressive than sporadic-IPF | 12-months of entering the study
  Disease progression defined as relative FVC decline ≥10% or death/lung transplant within 12 months of entering the study.

SECONDARY OUTCOMES:
All-cause mortality | Time of censoring or 12 months
Identify genotypes present in our study population | Within first 6 months of study recruitment
  Identify pathogenic genetic variants known to cause ILD present in our study population as well as at risk alleles e.g. MUC5B.
Change in quality of life scores from baseline to 1 year | From date of study entry (baseline) until 12-month-assessment questionnaire completed, 12 months
  Identify the number of participants with a change in their quality of life (QOL) scores over a twelve month period and if the change in QOL score is more likely to be associated factors such as genotype. Quality of life will be assessed based on the results of quality of life questionnaires completed including the Medical Research Council Dyspnoea Scale, Leicester Cough Questionnaire, The King's Brief Interstitial Lung Disease and EQ-5D-5L. The CTD-ILD cohort will also have Patient Global Assessment and Clinician Global Assessment scores recorded. These will be completed as close as possible to 0 months for the baseline score and at 6 and 12 months to assess for a change.
Change in 6MWT from baseline to 1 year | On entry to study (baseline) to end of observation period (12 months)
  6-Minute walk tests will be carried out in a clinical setting by a trained physiotherapist at baseline (0), 6 and 12 months.
Change in pulmonary function tests from baseline to 1 year | Baseline (0 months) to 12 month follow-up
  Changes in forced vital capacity and diffusing capacity of the lungs for carbon monoxide will be assessed
Changes and patterns in at home-spirometry with the patientMpower App | 12 Months
  Using the patientMpower App patients will take twice-weekly home spirometry readings which will be analysed for changes and patterns in spirometry readings
Change in HRCT scan | 12 months
  Comparison between baseline CT Thorax and follow-up CT scan 1 year later using American Thoracic Society Guidelines to determine if there is radiological progression.
Identify radiological phenotypes linked to disease behavior in pulmonary fibrosis | 12 months
  Use of computational methods to identify novel radiologic phenotypes linked to disease behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Killian Hurley, Principal Investigator — RCSI
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peljto AL, Blumhagen RZ, Walts AD, Cardwell J, Powers J, Corte TJ, Dickinson JL, Glaspole I, Moodley YP, Vasakova MK, Bendstrup E, Davidsen JR, Borie R, Crestani B, Dieude P, Bonella F, Costabel U, Gudmundsson G, Donnelly SC, Egan J, Henry MT, Keane MP, Kennedy MP, McCarthy C, McElroy AN, Olaniyi JA, O'Reilly KMA, Richeldi L, Leone PM, Poletti V, Puppo F, Tomassetti S, Luzzi V, Kokturk N, Mogulkoc N, Fiddler CA, Hirani N, Jenkins RG, Maher TM, Molyneaux PL, Parfrey H, Braybrooke R, Blackwell TS, Jackson PD, Nathan SD, Porteous MK, Brown KK, Christie JD, Collard HR, Eickelberg O, Foster EE, Gibson KF, Glassberg M, Kass DJ, Kropski JA, Lederer D, Linderholm AL, Loyd J, Mathai SK, Montesi SB, Noth I, Oldham JM, Palmisciano AJ, Reichner CA, Rojas M, Roman J, Schluger N, Shea BS, Swigris JJ, Wolters PJ, Zhang Y, Prele CMA, Enghelmayer JI, Otaola M, Ryerson CJ, Salinas M, Sterclova M, Gebremariam TH, Myllarniemi M, Carbone RG, Furusawa H, Hirose M, Inoue Y, Miyazaki Y, Ohta K, Ohta S, Okamoto T, Kim DS, Pardo A, Selman M, Aranda AU, Park MS, Park JS, Song JW, Molina-Molina M, Planas-Cerezales L, Westergren-Thorsson G, Smith AV, Manichaikul AW, Kim JS, Rich SS, Oelsner EC, Barr RG, Rotter JI, Dupuis J, O'Connor G, Vasan RS, Cho MH, Silverman EK, Schwarz MI, Steele MP, Lee JS, Yang IV, Fingerlin TE, Schwartz DA. Idiopathic Pulmonary Fibrosis Is Associated with Common Genetic Variants and Limited Rare Variants. Am J Respir Crit Care Med. 2023 May 1;207(9):1194-1202. doi: 10.1164/rccm.202207-1331OC. PMID 36602845
- [Background] Zhang D, Newton CA. Familial Pulmonary Fibrosis: Genetic Features and Clinical Implications. Chest. 2021 Nov;160(5):1764-1773. doi: 10.1016/j.chest.2021.06.037. Epub 2021 Jun 26. PMID 34186035
- [Background] Cutting CC, Bowman WS, Dao N, Pugashetti JV, Garcia CK, Oldham JM, Newton CA. Family History of Pulmonary Fibrosis Predicts Worse Survival in Patients With Interstitial Lung Disease. Chest. 2021 May;159(5):1913-1921. doi: 10.1016/j.chest.2021.01.026. Epub 2021 Jan 21. PMID 33484728
- [Background] Borie R, Kannengiesser C, Hirschi S, Le Pavec J, Mal H, Bergot E, Jouneau S, Naccache JM, Revy P, Boutboul D, Peffault de la Tour R, Wemeau-Stervinou L, Philit F, Cordier JF, Thabut G, Crestani B, Cottin V; Groupe d'Etudes et de Recherche sur les Maladies "Orphelines" Pulmonaires (GERM"O"P). Severe hematologic complications after lung transplantation in patients with telomerase complex mutations. J Heart Lung Transplant. 2015 Apr;34(4):538-46. doi: 10.1016/j.healun.2014.11.010. Epub 2014 Nov 13. PMID 25612863
- [Background] Tyndall AJ, Bannert B, Vonk M, Airo P, Cozzi F, Carreira PE, Bancel DF, Allanore Y, Muller-Ladner U, Distler O, Iannone F, Pellerito R, Pileckyte M, Miniati I, Ananieva L, Gurman AB, Damjanov N, Mueller A, Valentini G, Riemekasten G, Tikly M, Hummers L, Henriques MJ, Caramaschi P, Scheja A, Rozman B, Ton E, Kumanovics G, Coleiro B, Feierl E, Szucs G, Von Muhlen CA, Riccieri V, Novak S, Chizzolini C, Kotulska A, Denton C, Coelho PC, Kotter I, Simsek I, de la Pena Lefebvre PG, Hachulla E, Seibold JR, Rednic S, Stork J, Morovic-Vergles J, Walker UA. Causes and risk factors for death in systemic sclerosis: a study from the EULAR Scleroderma Trials and Research (EUSTAR) database. Ann Rheum Dis. 2010 Oct;69(10):1809-15. doi: 10.1136/ard.2009.114264. Epub 2010 Jun 15. PMID 20551155
- [Background] Navaratnam V, Fleming KM, West J, Smith CJ, Jenkins RG, Fogarty A, Hubbard RB. The rising incidence of idiopathic pulmonary fibrosis in the U.K. Thorax. 2011 Jun;66(6):462-7. doi: 10.1136/thx.2010.148031. Epub 2011 Apr 27. PMID 21525528
- [Background] Distler O, Highland KB, Gahlemann M, Azuma A, Fischer A, Mayes MD, Raghu G, Sauter W, Girard M, Alves M, Clerisme-Beaty E, Stowasser S, Tetzlaff K, Kuwana M, Maher TM; SENSCIS Trial Investigators. Nintedanib for Systemic Sclerosis-Associated Interstitial Lung Disease. N Engl J Med. 2019 Jun 27;380(26):2518-2528. doi: 10.1056/NEJMoa1903076. Epub 2019 May 20. PMID 31112379
- [Background] Yang M, Wu Y, Liu X, Zhao C, Li T, Li T, Zhang X, Jiang H, Mao B, Liu W. Efficacy and safety of antifibrotic agents in the treatment of CTD-ILD and RA-ILD: A systematic review and meta-analysis. Respir Med. 2023 Sep;216:107329. doi: 10.1016/j.rmed.2023.107329. Epub 2023 Jun 12. PMID 37315742